CLINICAL TRIAL: NCT04099433
Title: HPVinHIV: Study of Anal HPV Infection in the Setting of HIV Infected Individuals
Brief Title: Application of Oral Bacteriotherapy to Promote Anal HPV Clearance in HIV Positive Individuals
Acronym: HPVinHIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Prof. Gabriella d'Ettorre, Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4590
Record Dates: First submitted 2019-06-24; First posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: HIV; Anal Dysplasia
Keywords: HIV; HPV; Probiotics; High Resolution Anoscopy; Anal dysplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Bacteriotherapy Arm (Experimental): Individuals in this study arm will undergo 6 months of daily intake of an oral probiotic formulation (Vivomixx: 4 sachets/day, each sachet containing 450 billion live bacteria). Probiotic sachets are indistinguishable from placebo
  Interventions: Dietary Supplement: Vivomixx
- Placebo Arm (Placebo Comparator): Individuals in this study arm will undergo 6 months of daily intake of placebo (4 sachets/day). Placebo sachets are indistinguishable from probiotic
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vivomixx — Individuals in the interventional arm will undergo daily oral intake of probiotic supplement
  Arms: Oral Bacteriotherapy Arm
Other: Placebo — Individuals in the placebo arm will undergo daily oral intake of placebo supplement
  Arms: Placebo Arm

SUMMARY:
Published studies suggest that oral probiotic intake can promote the clearance of HPV genital infection and HPV related genital dysplasia in HIV negative women. In the present randomized, double blind, placebo controlled study, investigators will evaluate the ability of oral bacterio-therapy to enhance the clearance of anal HPV infection and anal HPV related dysplasia in HIV infected subjects.

Participants will be evaluated for anal HPV infection and anal dysplasia before and after a 6 months course of daily investigational product intake (Viviomixx® or placebo). HPV infection rate and presence of dysplasia at baseline and at the end of the study will be compared.

DETAILED DESCRIPTION:
Squamous Cell Carcinoma (SCC) of the anus and the anal canal represents a major concern for the HIV infected population, with incidence rates in the different sub populations (women, men, MSM) that are grater than those observed for other common neoplasms in the same HIV negative sub-populations. Nowadays, screening for anal precancerous dysplasia has been included in most national and international HIV management guidelines; in particular, italian guidelines suggest to screen for the presence of HPV related dysplasia:

* HIV+ MSM
* All individuals with previous or current evidence of ant-genital condyloma
* Women with cytology abnormalities on cervical Pap-smear Since no direct anti-HPV drug is currently available and control or clearance of the infection is possible only trough the effect of immune response, interest is addressed to find strategies to promote spontaneous clearance of infection.

In published studies, oral bacterio-therapy demonstrated the ability to promote HPV clearance and HPV related dysplasia regression in HIV negative women.

In the present randomized, double blind, placebo controlled trial, 40 HIV infected individuals with HPV related anal dysplasia will be enrolled.

At baseline participants will undergo:

* anal HPV research and identification
* anal cytology
* anal brushing for evaluation of local inflammatory milieu and microbiota

Subjects with identified HPV anal infection and anal dysplasia will undergo High Resolution Anoscopy (HRA).

During HRA, extra biopsies of identified abnormal areas and biopsies of normal mucosa will be obtained. Extra biopsies will be used to investigate the distribution of intra-epithelial immune cells populations.

Participants will then undergo 6 months of oral supplementation with probiotics (Vivomixx®) or placebo.

At the end of the supplementation period (Vivomixx or placebo), participants will undergo:

* anal HPV research and identification
* anal cytology
* anal brushing for evaluation of local inflammatory milieu and microbiota
* HRA

During HRA, extra biopsies of identified abnormal areas and biopsies of normal mucosa will be obtained. Extra biopsies will be used to investigate the distribution of intra-epithelial immune cells populations.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected individuals >18 years old
* stable and effective antiretroviral therapy since at least 12 months
* HPV associated anal dysplasia
* patient willing to provide written informed consent

Exclusion Criteria:

* impossibility to intake the investigational product
* any contraindication to blood sampling
* inflammatory bowel disease
* use of antibiotics during the 3 months prior to the enrollment in the study
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the number of HPV positive anal swabs | Anal swabs for HPV detection and genotyping will be performed at baseline and after the 6 months duration of the intervention
  Clearance of anal HPV infection will be defined as:
  * negative swab at the end of the study in participants with positive swab at baseline
  * positive swab at the end of the study that shows a different genotype from baseline
Change from baseline in the number of dysplastic lesions | Areas of the anal canal that were biopsied at baseline and whom histology showed the presence of dysplasia will undergo a second biopsy after the 6 months duration of the intervention
  Clearance of anal dysplasia will be defined as:
  - normal histology in biopsies repeated at the end of the study on areas that showed the presence of histologically defined dysplasia at baseline.

SECONDARY OUTCOMES:
Rate of adverse events | This measure will be assessed after the 6 months duration of the intervention
  The rate of adverse events occurred during the study period will be evaluated and compared between both groups
Comparison between intra-epithelial NK lymphocytes subpopulation in normal mucosa and dysplastic mucosa | Biopsies and intra-epithelial lymphocytes extraction will be performed at baseline and after the 6 months duration of the intervention
  Biopsies from dysplastic lesions and from normal mucosa will be taken at baseline. Biopsies will also be taken at the end of the study from previously biopsied areas, from normal mucosa and eventually from dysplastic areas that were not present at baseline. Intra-epithelial lymphocytes will be extracted from the biopsy tissue and stained to differentiate and quantify CD56+NK lymphocytes by flowcytometry. Changes from baseline will be expressed as relative difference.
Comparison between intra-epithelial CD4+ T lymphocytes subpopulation in normal mucosa and dysplastic mucosa | Biopsies and intra-epithelial lymphocytes extraction will be performed at baseline and after the 6 months duration of the intervention
  Biopsies from dysplastic lesions and from normal mucosa will be taken at baseline. Biopsies will also be taken at the end of the study from previously biopsied areas, from normal mucosa and eventually from dysplastic areas that were not present at baseline. Intra-epithelial lymphocytes will be extracted from the biopsy tissue and stained to differentiate and quantify CD4+ T lymphocytes by flowcytometry. Changes from baseline will be expressed as relative difference.
Comparison between intra-epithelial CD8+ T lymphocytes subpopulation in normal mucosa and dysplastic mucosa | Biopsies and intra-epithelial lymphocytes extraction will be performed at baseline and after the 6 months duration of the intervention
  Biopsies from dysplastic lesions and from normal mucosa will be taken at baseline. Biopsies will also be taken at the end of the study from previously biopsied areas, from normal mucosa and eventually from dysplastic areas that were not present at baseline. Intra-epithelial lymphocytes will be extracted from the biopsy tissue and stained to differentiate and quantify CD8+ T lymphocytes by flowcytometry. Changes from baseline will be expressed as relative difference.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pubblic Health and Infectious Diseases, "Sapienza" University of Rome, Rome, RM, Italy

REFERENCES:
- [Derived] Pedersen TB, Pachler FR, Rosenberg J, Andresen K. Interventions for anal canal intraepithelial neoplasia. Cochrane Database Syst Rev. 2025 Aug 13;8(8):CD009244. doi: 10.1002/14651858.CD009244.pub3. PMID 40801169